CLINICAL TRIAL: NCT04832074
Title: Immediate Stiffness Changes in Upper Trapezius Active Myofascial Trigger Points After Dry Needling in Patients With Neck Pain: A Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Immediate Stiffness Changes in Myofascial Trigger Points After Dry Needling
Acronym: ELECTROP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CamiloJcU21
Record Dates: First submitted 2021-03-30; First posted 2021-04-05 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2021-05

CONDITIONS: Myofascial Pain Syndrome; Neck Pain; Trigger Point Pain, Myofascial
MeSH Terms: conditions — Myofascial Pain Syndromes; Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blinded, Placebo-Controlled Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (Experimental): Dry needling will be performed with 'solid filiform needles'. The procedure is as follows: The participant will lie in the prone position. The overlying skin will be cleaned with antiseptic spray. The taut band and MTrP, will be localized manually.
  After measuring the Pain Pressure Thresholds in this location and the control (located 3 cm lateral to the MTrP), the needle within its plastic guide tube will be placed over the MTrP. After a tapping movement to insert the needle, the needle will be moved to the muscle around the bundle and moved forward and backward to the tissue to elicit a small muscle twitch. After eliciting LTR, needling will be stopped. If no twitch were elicited, needling will stopped after two or three stellate movements
  Interventions: Other: Dry Needling
- Sham Dry Needling (Sham Comparator): The same approach will be used with the exception of piercing the skin. The guide tube will press against the tissue and the sham needle will be allowed to drop against the skin. The handle will be tapped briskly but not breaking the skin. The sham needle will stay within the guide tube and will be pressed against the skin twice so as to mimic the quick "in and out" technique.
  Interventions: Other: Sham Dry Needling

INTERVENTIONS:
Other: Dry Needling — Real Dry Needling in the most active Myofascial Trigger Point
  Arms: Dry Needling
Other: Sham Dry Needling — Sham Dry Needling in the same location, but not piercing the skin
  Arms: Sham Dry Needling

SUMMARY:
Shear-wave elastography (SWE) is considered as a useful tool for quantifying muscle stiffness. Considering that Myofascial Trigger Points (MTrP) are defined as "hyperirritable zones in contracted bands of muscle, thought to be caused by muscle overload or stress" and the effectiveness of dry needling applied to active MTrP for reducing pain and disability, the aim of this study is to assess the effects of sham and real dry needling, applied to active MTrP in the upper trapezius muscle in patients with chronic neck pain, on the muscle stiffness in two areas: 1) the most symptomatic area and 2) a control point.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 and
* Presence of mechanical neck pain for at least three months duration
* Presence of at least one active MTrP in the Upper Trapezius muscle

Exclusion Criteria:

* Neck pain of traumatic origin (such as whiplash-associated disorder)
* Current use of any kind of analgesic therapy
* Presenting any condition usually considered a perpetuating factor of MTrPs, such as fibromyalgia, hypothyroidism, or iron deficiencies
* Presenting any contraindication for Dry Needling application
* Neuropathies (e.g., radiculopathy)
* Bilateral Pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
SWE - Young modulus | Baseline
  KPa
SWE - Young modulus | 10 minutes
  KPa
SWE - Local shear wave speed | Baseline
  m/s
SWE - Local shear wave speed | 10 minutes
  m/s
Pain Pressure Thresholds | Baseline
  kg/cm2
Pain Pressure Thresholds | 10 minutes
  kg/cm2

SECONDARY OUTCOMES:
Visual Analogue Scale | Baseline
  0-10
Neck Disability Index | Baseline
  0-100

CONTACTS AND LOCATIONS:
Overall Officials: Juan Antonio Valera-Calero, PhD, Principal Investigator — Camilo José Cela University
Locations (1):
- Francisco de Vitoria University, Pozuelo de Alarcón, Madrid, Spain

REFERENCES:
- [Derived] Valera-Calero JA, Sanchez-Jorge S, Buffet-Garcia J, Varol U, Fernandez-de-Las-Penas C, Alvarez-Gonzalez J. Changes in stiffness at active myofascial trigger points of the upper trapezius after dry needling in patients with chronic neck pain: a randomized controlled trial. Acupunct Med. 2023 Jun;41(3):121-129. doi: 10.1177/09645284221104831. Epub 2022 Jun 28. PMID 35765779